CLINICAL TRIAL: NCT03142438
Title: The Evaluation of a Full Face and Nasal Mask for the Treatment of Obstructive Sleep Apnea
Brief Title: The Evaluation of a Mask for the Treatment of Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Collaborators: North Texas Lung & Sleep Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIA-207
Record Dates: First submitted 2017-04-23; First posted 2017-05-05 (Actual); Results first posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-06

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- F&P Seal Improvement Project (Experimental): participants will be placed on this arm for a total of 14 +- 4 days from visit 1. participants will be using the trial mask during this treatment arm
  Interventions: Device: F&P Seal Improvement Project

INTERVENTIONS:
Device: F&P Seal Improvement Project — Participants will be placed on this arm for a total 14 ± 4 days from Visit 1. Participants will be using the trial full face or nasal mask during this treatment arm.

SUMMARY:
This investigation is a prospective, non randomized, non blinded study. This investigation is designed to evaluate the performance, comfort and ease of use with the F&P trial full face and nasal mask amongst Obstructive Sleep Apnea (OSA) patients. Up to 70 OSA patients will be recruited from the North Texas Lung and Sleep Clinic (NTLSC) database

DETAILED DESCRIPTION:
Visit 1 will involve the participants being fitted with the F&P trial full face or nasal mask for use in-home.

The participant will then come in to return the mask (Visit Two) and have a final interview, this ensures the maximum time participants will be exposed to the trial mask in home will be 14 ± 4 days from visit one.

The mask will be returned to the Institution at the conclusion of the trial and the participant will return to their previous mask. The Institution will recruit all patients within three weeks of the beginning of the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult (22+ years of age)
* Able to give informed consent
* Apnea hypopnea Index (AHI) ≥ 5 on diagnostic night
* Either prescribed Automatic positive airway pressure (APAP), Continuous positive airway pressure (CPAP) or Bi-level positive airway pressure (PAP) for OSA
* Fluent in spoken and written English
* Existing oronasal and nasal mask user

Exclusion Criteria:

* Inability to give informed consent
* Participant intolerant to PAP
* Anatomical or physiological conditions making PAP therapy inappropriate
* Current diagnosis of respiratory disease or carbon Dioxide (CO2) retention
* Pregnant or may think they are pregnant.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2017-06-23 (Actual); Study Completion 2017-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Ostransky, MD, Principal Investigator — Board Certified Sleep Specialist
Locations (1):
- North texas Lung and Sleep Clinic, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Investigation to inform product development team. Results will inform product development on the future of the product.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | F&P Seal Improvement Project
Started | 57
Completed | 57
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | F&P Seal Improvement Project
Number analyzed (Participants) | 57
Age, Customized [Count of Participants; unit: Participants]
  22 or older | 57
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 52
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 52
  New Zealand | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Subjective Usability Reporting
Description: Usability reported from participants questionnaires to evaluate the use of the F&P mask for treatment of Obstructive Sleep Apnea
Time Frame: 14 ± 4 days in-Home
Measure: Count of Participants; unit: Participants
Arm/Group | F&P Seal Improvement Project
Number analyzed (Participants) | 57
Participants
  Easier | 14
  The same | 41
  More difficult | 2

2. Primary Outcome: Number or Participants Comparative Subjective Reported Comfort
Description: Comfort reported from participants questionnaires to evaluate the use of the F&P mask for treatment of Obstructive Sleep Apnea compared to usual
Time Frame: 14 ± 4 days in-Home
Measure: Count of Participants; unit: Participants
Arm/Group | F&P Seal Improvement Project
Number analyzed (Participants) | 57
Participants
  More comfortable | 27
  The same | 24
  Less comfortable | 6

3. Secondary Outcome: Objective Performance Reporting
Description: Objective Apnea-Hypopnea Index (AHI) data recorded from the positive airway pressure (PAP) device to evaluate the use of the F&P mask for treatment of Obstructive Sleep Apnea
Time Frame: 14 ± 4 days in-Home
Measure: Count of Participants; unit: Participants
Arm/Group | F&P Seal Improvement Project
Number analyzed (Participants) | 57
Participants
  Lower AHI | 17
  No change in AHI | 3
  Higher AHI | 8
  Not collected | 29

4. Secondary Outcome: Number of Participants Reported Mask Acceptability
Description: Acceptability reported from participants questionnaires to evaluate the use of the F&P mask for treatment of Obstructive Sleep Apnea
Time Frame: 14 ± 4 days in-Home
Measure: Count of Participants; unit: Participants
Arm/Group | F&P Seal Improvement Project
Number analyzed (Participants) | 57
Participants
  Happy to use improved | 27
  Not happy to use improved | 18
  Happy to use either | 12

5. Secondary Outcome: Number of Participants Subjective Comfort Reporting
Description: Comfort reported from participants questionnaires to evaluate the use of the F&P mask for treatment of Obstructive Sleep Apnea
Time Frame: 14 ± 4 days in-Home
Measure: Count of Participants; unit: Participants
Arm/Group | F&P Seal Improvement Project
Number analyzed (Participants) | 57
Participants
  Very comfortable | 35
  Comfortable | 16
  Neither comfortable or uncomfortable | 4
  Uncomfortable | 2
  Very uncomfortable | 0

6. Secondary Outcome: Number or Participants Subjective Reporting of Seal Performance
Description: Seal performance reported from participants questionnaires to evaluate the use of the F&P mask for treatment of Obstructive Sleep Apnea
Time Frame: 14 ± 4 days in-Home
Measure: Count of Participants; unit: Participants
Arm/Group | F&P Seal Improvement Project
Number analyzed (Participants) | 57
Participants
  Very good | 28
  Good | 22
  Neither good nor poor | 6
  Poor | 1
  Very poor | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | F&P Seal Improvement Project
All-Cause Mortality (participants affected / at risk) | 0/57
Serious Adverse Events (participants affected / at risk) | 0/57
Other Adverse Events (participants affected / at risk) | 0/57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-12): https://cdn.clinicaltrials.gov/large-docs/38/NCT03142438/Prot_SAP_001.pdf